CLINICAL TRIAL: NCT02829502
Title: The Effect of Glucagon-like Peptide 1 (GLP-1) Receptor Agonist on Cerebral Blood Flow Velocity in Stroke Patients
Brief Title: The Effect of GLP-1 Receptor Agonist on Cerebral Blood Flow Velocity in Stroke
Acronym: EGRABIS1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christina Kruuse (Other)
Responsible Party: Sponsor-Investigator, Christina Kruuse, MD, PhD, DMSc, consultant Neurologist, Associate Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-16022538; 2016-001219-18 (EudraCT Number)
Record Dates: First submitted 2016-07-05; First posted 2016-07-12 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Ischemic Stroke
Keywords: Cerebrovascular disease; Glucagon like peptide 1
MeSH Terms: conditions — Ischemic Stroke; Cerebrovascular Disorders | interventions — Exenatide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Byetta (Active Comparator): Pre- and post treatment investigations:
  1. Mean flow velocity of the middle cerebral arteries bilateral by transcranial doppler
  2. Cerebral cortical oxygination by near infrared spectroscopy (NIRS)
  Endothelial function/response by the methods:
  * Biomarkers in blood (eg. e-selectin, VCAM, ICAM, endothelin, ADMA, miRNA)
  * EndoPAT2000
  * Ankle-brachial index
  Interventions: Drug: Byetta
- Normosaline (Placebo Comparator): Pre- and post treatment investigations:
  1. Mean flow velocity of the middle cerebral arteries bilateral by transcranial doppler
  2. Cerebral cortical oxygination by near infrared spectroscopy (NIRS)
  Endothelial function/response by the methods:
  * Biomarkers in blood (eg. e-selectin, VCAM, ICAM, endothelin, ADMA, miRNA)
  * EndoPAT2000
  * Ankle-brachial index
  Interventions: Drug: Normosaline

INTERVENTIONS:
Drug: Byetta — Single dose of subcutaneous injection of 5 μg exenatide (Byetta).
  Other Names: Exenatide; GLP-1 receptor analogue; GLP-1 receptor agonist
  Arms: Byetta
Drug: Normosaline — Single dose of subcutaneous injection of 20 μL normosaline (placebo).
  Other Names: Isotonic saline
  Arms: Normosaline

SUMMARY:
This randomized controlled trial investigates the effect of a single dose of glucagon-like peptide-1 (GLP-1) receptor agonist in the subacute phase of stroke in humans. The primary endpoint is the mean flow velocity in the middle cerebral arteries measured by transcranial doppler and cortical oxygination measured by near infrared spectroscopy (NIRS). The secondary endpoints are changes in endothelial/inflammatory biomarkers in the blood, changes in the ankle-brachial index and changes in the reactive hyperaemia index measured by EndoPAT2000.

DETAILED DESCRIPTION:
Glucagon-like peptide 1 (GLP-1) receptor agonists are widely used in the treatment of type 2 diabetes because of their ability to mimic the incretin hormone, GLP-1. GLP-1 increases glucose-dependent insulin secretion and thereby reduces the glucose level. Over the past few years, GLP-1 receptor agonists have been investigated as possible therapies for neurological disorders, due to their ability to cross the blood-brain-barrier. Evidence of the treatment of cerebrovascular diseases has been growing especially in animal stroke models. GLP-1 receptors, which are located in the central nervous system on neurons and endothelium, are upregulated in the brain due to ischemia. GLP-1 receptor agonists have shown anti-inflammatory and anti-apoptotic properties, and they may protect the cell from oxidative stress and may protect the endothelium. The inner lining of blood vessels, the endothelium, is an active component of the endocrine function. It affects the formation of blood clots and plays a role in the disease mechanisms of stroke. The current acute and prophylactic treatments of stroke mainly target platelet function, but not endothelial function.

This double-blinded, randomized, controlled, pilot trial investigates the effect of a single dose of the GLP-1 receptor agonist, exenatide, on cerebral blood flow velocity in the subacute phase of stroke in humans. The primary endpoint is the mean flow velocity in the middle cerebral arteries measured by transcranial doppler and cortical oxygination measured by near infrared spectroscopy (NIRS). The secondary endpoints are the effects on the peripheral endothelium, hereby: 1) changes in the reactive hyperaemia index measured by EndoPAT2000, 2) changes in the ankle-brachial index, and 3) changes in endothelial/inflammatory biomarkers in the blood. The primary and secondary endpoints are measured before and up till three hours after administration of exenatide.

The overall hypothesis is that GLP-1 receptor agonists may represent a novel potential neuroprotective treatment in stroke. Parallel to this study we investigate the effect of GLP-1 receptor agonist on people free of cerebrovascular diseases (ref. to EGRABINS1).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years with newly symptoms of stroke
* Able to receive exenatide/placebo within 21 days after onset of symptoms
* Radiological confirmed diagnoses of ischemic stroke
* NIHSS between 1-20 at the onset of symptoms
* modified rankin scale (mRS) ≤ 2 prior to onset of symptoms
* Has given written informed consent

Exclusion Criteria:

* Intracerebral haemorrhage
* Subdural / epidural hemorrhage
* Subarachnoid haemorrhage
* Previously major structural damage to the brain
* Diabetes type 1
* Diabetes type 2
* Known atrial fibrillation
* > 50% stenosis of internal carotid
* Known allergy to GLP-1 receptor agonists
* Hepatic impairment (ALT> 3 x upper normal limit)
* Renal impairment (eGFR <30 ml / min)
* Inflammatory bowel disease
* Previous pancreatitis
* Heart failure (NYHA class 3-4)
* Pregnancy or lactation
* Patient unable to co-operate to the investigation procedures
* Visualization of the middle cerebral artery bilaterally by transcranial dopple not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2023-08 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Changes in the mean flow velocity in the middle cerebral arteries and in cortical oxigination. | Up till 3 hours
  Change in the mean flow velocity in the middle cerebral arteries will be measured with transcranial doppler and cortical oxygination by near infrared spectroscopy (NIRS) before and up till tree hours after injection of exenatide/placebo.

SECONDARY OUTCOMES:
Endothelial reactivity | 3 hours
  Measurement of endothelial reactivity in fingers post occlusion by non-invasive plethysmography (EndoPAT2000) before and three hours after injection of exenatide/placebo.
Changes in endothelial biomarkers in blood | 3 hours
  Venous blood samples to measure endothelial biomarkers (including V-CAM, I-CAM, endothelin, e-selectin, ADMA, hsCRP, miRNA) before and three hours after injection of exenatide/placebo.
Endothelial function/response in ankle-brachial index | 3 hours
  Measuring of the blood pressure in the ankles and in the arm calculate the ankle-brachial index before and three hours after injection of exenatide/placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Christina R Kruuse, MD,PhD, Principal Investigator — Study Principal Investigator, Consultant Neurologist, Dept. Neurology, Herlev Hospital
Locations (1):
- Department of Neurology, Herlev-Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No